CLINICAL TRIAL: NCT06227013
Title: Promoting Whistleblowing Among Nurses: A Randomized Controlled Trail
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Port Said University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NUR (6/8/2023) (28)
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Nurse's Role
Keywords: Nurses; Whistleblowing
MeSH Terms: conditions — Whistleblowing

STUDY DESIGN:
Intervention Model Description: open-label, two-arm Randomized Control Trail (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): Whistleblowing intervention
  Interventions: Behavioral: Whistleblowing intervention
- control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Whistleblowing intervention — the participated nurses will receive session about Whistleblowing
  Arms: interventional group

SUMMARY:
this study aims to investigate the effect of Whistleblowing intension Among Nurses by applying whistobloating education program

DETAILED DESCRIPTION:
the study aims to assess the effectiveness of Whistleblowing intervention program on nurses'Whistleblowing intensions.

Hypotheses:

H1: Nurses participating in the Whistleblowing intervention will report, post intervention, high level of Whistleblowing intensions compared with those nurse nurses in control group

ELIGIBILITY:
Inclusion Criteria:

* licensed nurses who worked in direct contact with patients in their services had at least six month of experience in the nursing profession, agreed to participate in the study

Exclusion Criteria:

* participating in any intervention program within the last 12 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
easuring the change of the Whistleblowing intension of nurses | 3-months
  measuring changes occure in Whistleblowing intension after applied Whistleblowing programe yo nurses

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared to open data repository.
Supporting Information: Study Protocol
Time Frame: the data will be available after publishing the trail (expected in 2024)
Access Criteria: open access